CLINICAL TRIAL: NCT03757988
Title: Targeting Physical Health in Schizophrenia: Physical Activity Can Enhance Life
Acronym: PACE-life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-1296; 1R34MH111852-01A1 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Brief Psychotic Disorder; Schizophreniform Disorder; Unspecified Schizophrenia Spectrum and Other Psychotic Disorder
Keywords: Walking; Exercise; Physical Health
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Experimental Walking Group (Experimental): This is a pilot project with one single group that will be evaluated on the adherence to a walking protocol (Exercise Intervention- PACE-Life). Subjects will be walking two times a week under the supervision of the psychiatric clinic. In addition, subjects will be encouraged to add walking on their own on the days when subjects are not exercising under the supervision of the clinic. This pilot will be used to inform the final design of the subsequent randomized clinical trial that will be implemented following this pilot.
  Interventions: Behavioral: Exercise Intervention- PACE-Life

INTERVENTIONS:
Behavioral: Exercise Intervention- PACE-Life — Subjects will be provided with a Fitbit wristband and instructed how to use it. During the first group session, subjects will be taught how to use their heart rate (on the Fitbit) to determine how fast subjects should walk (to achieve the appropriate exercise dosage). Information on proper care, usage, and how to determine the appropriate heart rate from the watch, which will be used to guide the intensity of the walk will be provided to subjects and reviewed at each group session. For all clinic based group sessions, subjects will arrive at the STEP clinic to meet the entire group and leaders and be reminded of the HR that corresponds with the intensity of that group session. Next, the group will go outside and walk for 30 minutes.

SUMMARY:
Purpose: To develop and test the feasibility of an exercise intervention that combines group walking, activity tracking, and heart rate monitoring, and determine the effectiveness of this intervention on the physical and mental health for individuals with schizophrenia spectrum disorders.

Participants: 14 individuals with schizophrenia spectrum disorders.

Procedures (methods): During the baseline assessment, subjects will be provided with a Fitbit wristband and instructed how to use it. During the first group session, subjects will be taught how to use their heart rate (on the Fitbit) to determine how fast subjects should walk (to achieve the appropriate exercise dosage). Information on proper care, usage, and how to determine the appropriate heart from the watch, which will be used to guide the intensity of the walk will be provided to subjects and reviewed at each group session. For all clinic based group sessions, subjects will arrive at the STEP clinic to meet the entire group and leaders and be reminded of the heart rate (HR) that corresponds with the intensity of that group session. Next, the group will go outside and walk for 30 minutes. At the completion of 30 minutes, everyone will go back into the clinic for water and review of the walk. After the second group session of each week, subjects will receive weekly progress reports of their steps and minutes spent walking the prior week (obtained from Fitbit devices). During this session, subjects will also set individual goals for the upcoming week for both their "intensity walks" and total steps per day.

DETAILED DESCRIPTION:
Overview of Procedures: PACE-life will be integrated into the Schizophrenia Treatment and Evaluation Program (STEP) outpatient clinics in Raleigh, NC and Carrboro, NC. The group walks will occur in the surrounding area around the clinics on sidewalks, bike trails, and residential streets. Goal setting groups and all assessments will take place in a conference room at the clinic. Goal-setting will include setting goals for the upcoming week in terms of number of steps as well as how many intensity walks that individuals plan to complete.

Assessments/Measures: The exercise intervention, PACE-Life, will last for 24 weeks and includes both group walks and independent walks (done at a location of the subject's choosing). Participants will be asked to complete assessments at screening, baseline, mid-point, post-test, and 1-month follow-up (approximately 28 weeks total).

At Screening the following measures will be examined: Demographics, the Wechsler Abbreviated Scale of Intelligence (WASI), a licensed physician will complete a medical history and physical exam, Physical Activity Readiness Questionnaire (PAR-Q).

At Baseline, Mid-point, Post-test, and 1-Month Follow-up the following measures will be examined: Demographics, Minutes Spent Walking, the Short Form International Physical Activity Questionnaire (IPAQ), Steps/day, Cardiorespiratory fitness (CRF)- CRF will be measured using the 6-minute walk test (6MWT), Self-determination Basic Needs, the Basic Psychological Need Scale-in General, the Basic Psychological Needs in Exercise Scale (BPNES), the Mini International Neuropsychiatric Interview (MINI) (Baseline Only), Resting Systolic/Diastolic Blood Pressure and resting heart rate (RHR), autonomous motivation will be measured with the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2), enjoyment of walking will be measured with the Physical Activity Enjoyment Scale (PACES), the UCLA Loneliness Scale, Weight, BMI, and Waist/hip Circumference.

At the conclusion of the open trial, the investigators will administer a brief questionnaire to the subjects regarding satisfaction and acceptability that will have both forced choice and open-ended questions.

Intervention- Groups will occur twice per week for 30 minutes for the entire intervention without changes in frequency and duration. The intensity, however, of both group walks and home-based walks will increase throughout this intervention in a stepwise fashion to create an exercise dose response to maximize impact on CRF.

Fitbits: All participants will be provided a Fitbit that is labeled with a participant number. All Fitbits are paired to a Fitbit account. Data from Fitbit devices can be synced to the corresponding account and accessed through Fitbit.com. Participants will be provided information about their accounts should participants want to look at the data but will be asked not to change any of the settings as the investigators will be using data for tracking steps/day and minutes spent walking.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) diagnosis of a Schizophrenia Spectrum Disorder (SSD) (Schizophrenia, Schizoaffective Disorder, Brief Psychotic Disorder, Schizophreniform Disorder, and Unspecified Schizophrenia Spectrum and Other Psychotic Disorder)
* Between the ages of 18-65, both genders, and any ancestry;
* Intelligence Quotient (IQ) >70. IQ will be assessed using the WASI
* No hospitalizations for psychiatric reasons in the last 3 months
* Clinically stable (no psychiatric medication changes within the past month)
* Are not already engaging in consistent moderate-intensity exercise (cutoff = 60 min/week for the past 6 months);
* Present with no contra-indication to engage in regular moderate intensity exercise based on the American College of Sports Medicine guidelines. (If an individual answers yes to one item on the of the Physical Activity Readiness Questionnaire (PAR-Q), a questionnaire that assesses cardiovascular risk factors, she/he will be asked to get clearance from a physician prior to participating in the study)
* Willing and able to provide informed consent. (Note: The research assistant will read the consent form with the participant and ask the subject to repeat back the information after each section to determine whether he/she understands the information provided.)

Exclusion Criteria:

* Pregnant women will be excluded because pregnancy alters autonomic and immune responsiveness, increase weight gain, and can influence heart rate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Penn, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - North Carolina Psychiatric Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months following publication
Access Criteria: Requesting investigator has appropriate approval (see above) and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Experimental Walking Group: This is a pilot project with one single group that will be evaluated on the adherence to a walking protocol (Exercise Intervention- PACE-Life). Subjects will be walking two times a week under the supervision of the psychiatric clinic. In addition, subjects will be encouraged to add walking on their own on the days when subjects are not exercising under the supervision of the clinic. This pilot will be used to inform the final design of the subsequent randomized clinical trial that will be implemented following this pilot.
  Exercise Intervention- PACE-Life: Subjects will be provided with a Fitbit wristband and instructed how to use it.
Period: Overall Study
Arm/Group | Single Arm Experimental Walking Group
Started | 17
Completed | 16
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.188 (11.743)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Pacific Islander | 2
  Black or African American | 3
  White | 9
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Participant's Total Distance During 6-Minute Walk From Baseline to Week 24
Description: The 6-minute walk test (6MWT) will be used to measure cardiorespiratory fitness (CRF) during which individuals will be asked to walk continuously for six minutes on a flat, indoor surface around cones (separated by 100 ft). The possible distance range is 400 meters to 650 meters. Higher scores reflect better outcomes (greater physical fitness).
Time Frame: Baseline, Post Treatment (24 weeks)
Population: Includes participants with data at Baseline and Post Treatment
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
meters | 92.420 (95.490)

2. Primary Outcome: Mean Difference in Participant's Total Distance During 6-Minute Walk From Post Treatment to Week 28
Description: as for outcome 1
Time Frame: Post Treatment (24 weeks), Follow-Up (Up to 28 weeks)
Population: Includes participants with data at Post Treatment and Follow-Up
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 8
meters | 6.65 (32.599)

3. Secondary Outcome: Mean Difference Overall UCLA Loneliness Scale Score
Description: Mean difference in overall score from Baseline to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). The UCLA Loneliness scale is a 20 item scale. Answers are on a 4 point scale with options "I often feel this way," "I sometimes feel this way," "I rarely feel this way," and "I never feel this way." Possible scores range from 20 to 80. Higher scores reflect worse outcomes (greater feelings of loneliness).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
score on a scale
  Baseline to Post Treatment | 0.133 (9.172)
  Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Post Treatment to Follow-Up | -1.778 (8.511)

4. Secondary Outcome: Mean Difference Overall PANSS Score
Description: Mean difference in the overall score from Baseline to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). The PANSS is a semi-structured interview using a 30-item scale to evaluate the presence, absence and severity of Positive, Negative and General Psychopathology symptoms of schizophrenia. All 30 items are rated on a 7-point scale (1 = absent; 7 = extreme). Possible scores range from 30 to 210. Higher scores reflect worse outcomes (i.e. greater symptoms of psychosis).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
score on a scale
  Baseline to Post Treatment | 8.267 (12.151)
  Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Post Treatment to Follow-Up | -2.778 (7.661)

5. Secondary Outcome: Mean Difference in Body Mass Index (BMI)
Description: Mean difference in body mass index (BMI) from Baseline to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). Higher scores reflect worse outcomes (i.e. greater body mass).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
kg/m^2
  Baseline to Post Treatment | 0.280 (1.736)
  Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Post Treatment to Follow-Up | 0.022 (0.640)

6. Secondary Outcome: Mean Difference in Diastolic Blood Pressure Change
Description: Mean difference in diastolic blood pressure change from Baseline to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). Normal diastolic blood pressure ranges from ≤ 70 to higher than 120 mmHg. Higher scores reflect worse outcomes (i.e., higher diastolic blood pressure).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
mmHg
  Baseline to Post Treatment | 5.667 (12.675)
  Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Post Treatment to Follow-Up | 5.333 (7.566)

7. Secondary Outcome: Mean Difference in Systolic Blood Pressure Change
Description: Mean difference in systolic blood pressure change from Baseline to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). Normal systolic blood pressure ranges from ≤120 to higher than 140 mmHg. Higher scores reflect worse outcomes (i.e., higher systolic blood pressure).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
mmHg
  Baseline to Post Treatment | 1.733 (10.402)
  Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Post Treatment to Follow-Up | 11.111 (13.110)

8. Secondary Outcome: Mean Difference in Resting Heart Rate Change
Description: Mean difference in resting heart rate change from Baseline to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). Normal heart rate ranges from ≤ 60 to higher than 100. Higher scores reflect worse outcomes (poorer heart condition).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
beats per minute
  Baseline to Post Treatment | 1.533 (19.460)
  Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Post Treatment to Follow-Up | 2.667 (13.115)

9. Secondary Outcome: Mean Difference in Waist Circumference
Description: Mean difference in waist circumference from Baseline to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). Normal waist circumference ranges ≤ than 94cm for males and < than 80 for females to higher than 102 cm for males and 88cm for females . Higher scores reflect worse outcomes (i.e. greater waist circumference = disease development risk).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
centimeters
  Baseline to Post Treatment | 2.533 (9.226)
  Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Post Treatment to Follow-Up | -0.667 (2.411)

10. Secondary Outcome: Mean Difference in Weight
Description: Mean difference in weight from Baseline to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). Normal weight ranges from 45 to 130 kilograms . Higher scores reflect worse outcomes (i.e., greater weight).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
kilograms
  Baseline to Post Treatment | 0.887 (4.659)
  Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Post Treatment to Follow-Up | 0.556 (1.384)

11. Other Pre Specified Outcome: Mean Difference in Weighted Average Motivation Score (Relative Autonomy Index) on the Behavioral Regulation Exercise Questionnaire (BREQ-2)
Description: Mean difference in weighted average motivation score (relative autonomy index) from Baseline to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). The BREQ-2 is a 19 item self-report scale. Answers are on a 5 point Likert scale ranging from 0 to 4. Zero corresponds to "not true for me" and 4 corresponds to "very true for me." Possible scores range from -24 to +20. Each subscale is calculated from averages (items scored 0-4) and then a weight is applied. Higher scores reflect better outcomes (higher autonomous motivation to exercise).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
score on a scale
  Baseline to Post Treatment | -0.906 (5.476)
  Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Post Treatment to Follow-Up | 0.157 (2.379)

12. Other Pre Specified Outcome: Mean Difference in Subscale Scores on the Basic Psychological Needs in Exercise Scale (BPNE)
Description: Mean difference in subscale scores of autonomy, relatedness, and competence from Baseline to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). The BPNE is an 11 item self-report scale. Answers are on a 5 point Likert scale ranging from "I don't agree at all" to "I completely agree." Possible scores for each subscale range from 1 to 5. Higher scores reflect better outcomes (i.e. more psychological needs being met through exercise).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
score on a scale
  Autonomy scores from Baseline to Post Treatment | 0.383 (0.944)
  Relatedness scores from Baseline to Post Treatment | 0.978 (1.483)
  Competence scores from Baseline to Post Treatment | 0.250 (1.225)
  Autonomy scores from Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Autonomy scores from Post Treatment to Follow-Up | -0.222 (0.491)
  Relatedness scores fromPost Treatment to Follow-Up: number analyzed (Participants) | 9
  Relatedness scores fromPost Treatment to Follow-Up | -0.333 (1.080)
  Competence scores from Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Competence scores from Post Treatment to Follow-Up | -0.194 (0.873)

13. Other Pre Specified Outcome: Mean Difference in Subscale Scores on the Basic Psychological Need Scale - in General (BPNS)
Description: Mean difference in subscale scores of autonomy, relatedness, and competence from Baseline to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). 2. The BPNS is a 21-item self-report scale. Answers are on a 7 point Likert scale ranging from "Not at all true" to "Very true." Possible scores for each subscale range from 1 to 7. Higher scores reflect better outcomes (i.e more psychological needs being met).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
score on a scale
  Autonomy scores from Baseline to Post Treatment | 0.067 (1.132)
  Relatedness scores from Baseline to Post Treatment | 0.017 (0.836)
  Competence scores from Baseline to Post Treatment | 0.000 (0.970)
  Autonomy scores from Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Autonomy scores from Post Treatment to Follow-Up | 0.079 (1.050)
  Relatedness scores fromPost Treatment to Follow-Up: number analyzed (Participants) | 9
  Relatedness scores fromPost Treatment to Follow-Up | -0.152 (0.335)
  Competence scores from Post Treatment to Follow-Up: number analyzed (Participants) | 9
  Competence scores from Post Treatment to Follow-Up | -0.019 (0.709)

14. Other Pre Specified Outcome: Median Difference in Daily Steps From Fitbit Devices
Description: Median difference in steps/day from Week 1 to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). Fitbit devices record steps taken. Higher scores reflect better outcomes (higher steps/day).
Time Frame: Up to 28 weeks
Population: Includes participants with data at Baseline, Post Treatment, and Follow-Up. If estimate is missing for baseline or posttest, the closest point within three weeks was used as an estimate.
Measure: Median (Full Range); unit: steps per day
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
steps per day
  Week 1 to Post Treatment: number analyzed (Participants) | 7
  Week 1 to Post Treatment | -228 [-14752 to 3834]
  Post Treatment to Follow-Up: number analyzed (Participants) | 8
  Post Treatment to Follow-Up | -31.5 [-6223 to 4291]

15. Other Pre Specified Outcome: Median Difference in Minutes Spent Walking From Fitbit Devices
Description: Median difference in weekly minutes spent walking from Week 1 to Post Treatment (24 weeks) and to Follow-Up Visit (up to 28 weeks). Fitbit devices record minutes spent walking in bouts of 15 minutes. Higher scores reflect better outcomes (higher weekly minutes spent walking).
Time Frame: Up to 28 weeks
Population: as for outcome 14
Measure: Median (Full Range); unit: minutes per week
Arm/Group | Single Arm Experimental Walking Group
Number analyzed (Participants) | 15
minutes per week
  Week 1 to Post Treatment: number analyzed (Participants) | 7
  Week 1 to Post Treatment | -55.0 [-1571 to 8]
  Post Treatment to Follow-Up: number analyzed (Participants) | 8
  Post Treatment to Follow-Up | 27.5 [-78 to 108]

ADVERSE EVENTS:
Time Frame: From the time of Informed Consent through follow-up, up to approximately 28 weeks
Arm/Group | Single Arm Experimental Walking Group
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 3/17
Other Adverse Events (participants affected / at risk) | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Experimental Walking Group (N=17)
Psychiatric Hospitalization Due to Medication Non-Adherence (Psychiatric disorders) | 2 (2)
Psychiatric Hospitalization (Psychiatric disorders) | 1 (1)
Increased Psychiatric Symptoms (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03757988/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03757988/SAP_001.pdf